CLINICAL TRIAL: NCT00579826
Title: Study of Breast Cancer Prevention by Letrozole in High Risk Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: Novartis (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10587; CFEM345AUS45 (Other Grant/Funding Number: Novartis); 5R01CA122577-03 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Letrozole (Experimental): Letrozole, 2.5 mg daily for 6 months
  Interventions: Drug: Letrozole
- Placebo (Placebo Comparator): Placebo, daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg tablet daily. Then optional open label letrozole for another 6 months.
  Other Names: Letrozole(Femara)
  Arms: Letrozole
Drug: Placebo — Placebo tablet daily for 6 months then optional open label letrozole for 6 months.
  Arms: Placebo

SUMMARY:
This is a multi-institution double-blind placebo-controlled trial whose main objective is to determine if 6 months of letrozole (2.5 mg daily) can reduce proliferation as assessed by Ki-67 in high risk postmenopausal women on systemic hormone replacement therapy who have random periareolar fine needle aspiration (RPFNA) evidence of hyperplasia with atypia or borderline atypia, and a minimum Ki-67 of >1.5%.

The primary hypothesis is that proliferation and expression of other estrogen response genes will be favorably modulated by six months of letrozole relative to placebo without substantially increasing hot flashes or worsening overall quality of life.

DETAILED DESCRIPTION:
Subsequent to the 6 month RPFNA for assessment of biomarkers, toxicity and quality of life assessments, all women may receive optional open-label letrozole for an additional 6 months, followed by a third RPFNA and biomarker

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women at high risk for development of breast cancer
* stable dose of hormone replacement therapy
* have cytomorphologic evidence of hyperplasia +/- atypia and Ki-67 expression >1.5% in benign breast epithelial cells acquired by RPFNA
* Serum level of 25-hydroxyvitamin D of at least 30 ng/ml prior to study entry
* Willing to have a repeat random periareolar fine needle aspiration (RPFNA) and mammogram at 6 months and 12 months (if participating in the open label portion of the study) following initiation of study drug

Exclusion Criteria:

* Prior history of osteoporosis or osteoporotic fracture.
* Prior history of invasive breast cancer or other invasive cancer within five years from date of study entry.
* Current and chronic use of cyclooxygenase-2 (COX-2) specific inhibitors or NSAIDs
* Receiving treatment for rheumatoid arthritis or fibromyalgia
* Current history of poorly controlled migraines or perimenopausal symptoms
* Currently receiving other investigational agents.
* Receipt of more than 6 months of an aromatase inhibitor (anastrozole, exemestane, letrozole, etc.) at any time in the past.

Ages: 30 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-10; Primary Completion 2015-03 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Global results will be published.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Letrozole | Placebo
Started | 29 | 26
6 Months | 28 (RPFNA for assessment for primary endpoint.) | 25 (RPFNA for assessment for primary endpoint.)
Completed | 24 (Optional open label letrozole months 6-12; followed by RPFNA,) | 23 (Optional open label letrozole months 6-12; followed by RPFNA,)
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Population: All enrolled subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Letrozole | Placebo | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (8.3) | 44.7 (7.4) | 57.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 29 | 25 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 26 | 55
Height [Mean (Standard Deviation); unit: m] | 1.63 (0.09) | 1.64 (0.08) | 1.63 (0.08)
Weight [Mean (Standard Deviation); unit: kg] | 69.0 (11.2) | 73.6 (15.9) | 71.2 (13.7)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.0) | 27.9 (9.1) | 27.0 (7.2)
Age at menarche [Mean (Standard Deviation); unit: years] | 12.6 (1.3) | 12.6 (1.2) | 12.6 (1.2)
Age at first live birth [Mean (Standard Deviation); unit: years] | 20.5 (10.1) | 21.7 (11.1) | 21.4 (10.2)
History of prior breast biopsy [Number; unit: participants]
  History of biopsy | 19 | 16 | 35
  No history of biopsy | 10 | 10 | 20
History of prior Ductal Carcinoma In Situ (DCIS) or Lobular Carcinoma in Situ (LCIS) [Number; unit: participants]
  History | 3 | 1 | 4
  No History | 26 | 25 | 51
Number of relatives with breast cancer [Number; unit: participants]
  With relatives | 18 | 20 | 38
  No relatives | 11 | 6 | 17
Gail risk of developing breast cancer within 5 years [Mean (Standard Deviation); unit: percent] | 4.2 (3.9) | 3.4 (1.8) | 3.8 (3.1)
Immunocytochemical expression of Ki-67 [Mean (Standard Deviation); unit: percent] — Percent of breast epithelial cells staining positive for Ki-67 by immunocytochemistry.
  percent | 4.5 (3.1) | 4.0 (2.8) | 4.2 (3.0)
Cytology [Number; unit: participants]
  Hyperplasia | 4 | 4 | 8
  Hyperplasia with borderline atypia | 5 | 5 | 10
  Hyperplasia with Atypia | 20 | 17 | 37
Masood Score [Mean (Standard Deviation); unit: units on a scale] — Semi-quantitative cytology index score reflecting increasing abnormality, thus higher scores are worse. Range 6 to 24.
  units on a scale | 15 (0.9) | 15 (1.1) | 15 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Proliferation Rate (Ki-67 by Immunocytochemistry) From Baseline to 6 Months
Description: Change in proliferation rate (percent positively stained cells for Ki-67 antigen by immunocytochemistry) in benign breast epithelial cells acquired by random periareolar fine needle aspiration (RPFNA) from women at high risk for the development of breast cancer.
Time Frame: Baseline to 6 Months
Population: Subjects who complete initial 6-month period and have repeat RPFNA.
Measure: Mean (Standard Deviation); unit: percentage of cells stained positive
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 28 | 25
percentage of cells stained positive | -1.5 (2.8) | -1.1 (3.9)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.92, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Assessment of Change in Morphology by the Masood Score.
Description: Masood score is a semi-quantitative index of increasing abnormality, thus higher values are worse. Range 6 to 24.
  Based on Masood S, Frykberg ER, McLellan GL, Scalapino MC, Mitchum DG, Bullard JB. Prospective evaluation of radiologically directed fine-needle aspiration biopsy of nonpalpable breast lesions. Cancer 1990; 66:1480-7.
Time Frame: Baseline to 6 Months
Population: Subjects who complete initial 6-month intervention and have a repeat RPFNA, thus a change from baseline to 6-months can be computed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 28 | 25
units on a scale | -1.1 (1.5) | -1.1 (1.8)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.96, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Mammographic Density From Baseline to 6 Months..
Description: Percent area of the breast considered to be at increased density, as determined by the computer program Cumulus..
Time Frame: Baseline to 6 Months
Population: Subjects who complete the initial 6-months intervention and have mammograms available for analysis at baseline and 6 months, thus a change can be computed.
Measure: Mean (Standard Deviation); unit: percent of breast area at high density
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 23 | 24
percent of breast area at high density | -3.8 (12.8) | 0.2 (11.8)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority or Other; p = 0.73, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Change in Fibromyalgia Impact Questionnaire (FIQ) Score.
Description: Assessment of impact of fibromyalgia on everyday living activities. Composite score ranges from 0 (best, no interference or impact on activities) to 104 (worst, maximum interference with activities).
Time Frame: Baseline to 6 months
Population: subjects who complete 6 month visit and provide a 6-month FIQ score, such that the change in score (6-month - baseline) can be computed.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 25 | 24
score on scale | 3.7 (9.6) | 3.9 (10.3)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.64, Wilcoxon (Mann-Whitney)

5. Other Pre Specified Outcome: Change in Brief Fatigue Inventory (BFI) Score.
Description: Assessment of the extent to which fatigue interferes in normal everyday living activities. Change over 6 months of treatment is assessed. Range from 0 (best, no fatigue) to 10 (worst). Increase in score indicates greater intensity of fatigue and/or greater interference with activities due to fatigue.
Time Frame: baseline to 6 months
Population: Subjects who complete a 6-months visit and a 6-months BFI questionnaire, such that change in score can be computed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Letrozole | Placebo
Number analyzed (Participants) | 26 | 25
score on a scale | 0.6 (1.9) | 0.4 (1.6)
Statistical Analysis 1: Comparison: Letrozole vs Placebo; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: duration of study agent
Groups:
- Letrozole, 2.5 mg Daily for 12 Months: Letrozole, 2.5 mg daily for 6 months
  Letrozole: Letrozole 2.5 mg tablet daily. Then optional open label letrozole for another 6 months.
- Placebo for 6 Months; Open Label Letrozole 2.5 mg Daily: Placebo, daily for 6 months
  Placebo: Placebo tablet daily for 6 months then optional open label letrozole for 6 months.
Arm/Group | Letrozole, 2.5 mg Daily for 12 Months | Placebo for 6 Months; Open Label Letrozole 2.5 mg Daily
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 11/29 | 3/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letrozole, 2.5 mg Daily for 12 Months (N=29) | Placebo for 6 Months; Open Label Letrozole 2.5 mg Daily (N=26)
Cataract (Eye disorders) | 1 (2) | 0 (0) — Grade 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) — Grade 3
Atrial Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — Grade 3
Wound complication (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 3
Gallbladder necrosis (Hepatobiliary disorders) | 1 (1) | 0 (0) — Grade 3
Kidney pain (Renal and urinary disorders) | 0 (0) | 1 (1) — Grade 3
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) — Grade 3
Vomiting/nausea (Gastrointestinal disorders) | 1 (3) | 0 (0) — Grade 3
Headache (Nervous system disorders) | 1 (2) | 0 (0) — Grade 3
Vaginal mucositis/ cervical infection (Reproductive system and breast disorders) | 1 (2) | 0 (0) — Grade 3
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT00579826/Prot_SAP_000.pdf